CLINICAL TRIAL: NCT05424796
Title: Postoperative Pain Intensity Following Pulpotomy With Different Disinfection and Hemostatic Procedures in Teeth With Symptomatic Irreversible Pulpitis: a Randomized Clinical Trial
Brief Title: Postoperative Pain Intensity After Pulpotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Muhammed Ayhan, Research assistant, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cumhuriyet-University-M-AYHAN-
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Irreversible pulpitis; KTP laser; mineral trioxide aggregate; postoperative pain; pulpotomy; visual analog scale
MeSH Terms: conditions — Pain, Postoperative | interventions — Hemostasis; Lasers, Solid-State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Physiological saline (Control group) (n=30) (Experimental): In this group, hemostasis was achieved by checking the saline soaked cotton pellet placed over canal orifices and into the pulp chamber at 2-minute intervals.
  Interventions: Combination Product: Physiological saline
- Group 2: Hemostasis and cavity disinfection with NaOCl (n=30) (Experimental): In this group, 2.5% NaOCl soaked cotton pellets were placed over canal orifices and into the pulp chamber to achieve complete hemostasis.
  Interventions: Combination Product: Hemostasis and cavity disinfection with NaOCl
- Group 3: Hemostasis and cavity disinfection with KTP laser (n=30) (Experimental): In this group, complete hemostasis and cavity disinfection were achieved using a KTP laser (SMARLITE D, Deka, Calenzano FI, Italy). After initial hemorrhage control, complete hemostasis was achieved by exposure to a KTP laser (532 nm wavelength) in noncontact mode at 1.5 W of power with a pulse mode (Ton 100 ms, Toff 100 ms) for 2 s. The diameter of optical fiber was 300 μm. Laser application was repeated 3 times if required. After bleeding control was achieved, cavity disinfection was performed by laser application with a noncontact circular movement for 5 s using 1 W power and 300 nm tip.
  Interventions: Device: Hemostasis and cavity disinfection with KTP laser

INTERVENTIONS:
Combination Product: Physiological saline — Pulpotomy is a vital pulp treatment in which the vital coronal pulp tissue is surgically removed and the remaining radicular dental pulp is covered with an appropriate material. In this group, hemostasis was achieved by checking the saline soaked cotton pellet.
  Arms: Group 1: Physiological saline (Control group) (n=30)
Combination Product: Hemostasis and cavity disinfection with NaOCl — Pulpotomy is a vital pulp treatment in which the vital coronal pulp tissue is surgically removed and the remaining radicular dental pulp is covered with an appropriate material. In this group, 2.5% NaOCl soaked cotton pellets were placed over canal orifices.
  Arms: Group 2: Hemostasis and cavity disinfection with NaOCl (n=30)
Device: Hemostasis and cavity disinfection with KTP laser — Pulpotomy is a vital pulp treatment in which the vital coronal pulp tissue is surgically removed and the remaining radicular dental pulp is covered with an appropriate material. In this group, complete hemostasis and cavity disinfection were achieved using a KTP laser (SMARLITE D, Deka, Calenzano FI, Italy).
  Arms: Group 3: Hemostasis and cavity disinfection with KTP laser (n=30)

SUMMARY:
Introduction: This study aimed to compare postoperative pain rates following sodium hypochlorite (NaOCl) and KTP laser-assisted pulpotomy treatments in permanent teeth with deep caries, and symptomatic irreversible pulpitis. Methods: Ninety patients complaining of permanent teeth pain due to symptomatic irreversible pulpitis were randomly divided into 3 equal groups. Preoperative pain levels were recorded. After the initial bleeding control was achieved with saline, complete hemostasis was achieved by applying saline (control group), 2.5% NaOCl, or KTP laser according to randomly determined patient groups. Patients were asked to mark their pain level on the visual pain scale at the 6th, 24th, 48th, and 72nd hours, and 7th and 30th days depending on the severity of the pain. The permanent restoration was completed after 7 days. Results: According to the present study, the statistical difference between the groups in terms of preoperative pain and percussion pain levels was insignificant.

There was no significant difference between the groups in terms of demographic data. The postoperative pain level of the KTP laser group was significantly lower at the 6th hour compared to the saline group. There was no significant difference between the groups in terms of postoperative pain level at other time intervals. The greatest pain scores occurred in all groups at 6th hour. Conclusions: KTP laser can be preferred primarily in reducing postoperative pain in pulpotomy treatments. KTP laser or NaOCl assisted pulpotomy can be an effective treatment for pain reduction in permanent teeth with symptomatic irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be ≥ 18 years old, a single tooth in every patient
* Must be signs of irreversible pulpitis, such as persistent pain that begins spontaneously and/or is exacerbated by cold. This situation should be repeated with the cold test.
* Irreversible pulpitis diagnosed, with or without symptomatic apical periodontitis
* No systemic disease
* Should give a positive response to electrical and thermal tests
* Must be the opposite tooth.
* The tooth is restorable, probing pocket (3mm) depth, and mobility are within normal limits

Exclusion Criteria:

* Presence of allergies
* Using analgesics in the last 12 hours or antibiotics in the last 1 week before the procedure.
* Presence of swelling, palpation pain or sinus tract before treatment, root fracture or crack.
* Failure to control bleeding within 6 minutes,
* Presence of bruxism or open apex.
* Insufficient bleeding after pulp exposure
* Observation of advanced canal calcification
* Presence of internal or external root resorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity on the visual analog scale (VAS) at 6, 24, 48, and 72 hours, and 7 and 30 days after treatment. | Baseline and at 6, 24, 48 and 72 hours, and 7 and 30 days after treatment.
  The preoperative pain values of the patient were marked on the visual analog scale by the patient. The intensity of the pain was calculated by measuring the area in which the individual was marked between 0 (no pain) and 100 (worst pain). Patients recorded postoperative pain levels on the VAS for pain from 0 (no pain) to 100 (worst pain) at 6, 24, and 48 hours, and 7 and 30 days after treatment.

SECONDARY OUTCOMES:
Change from baseline in percussion values on the visual analog scale (VAS) at 7 and 30 days after treatment. | Baseline and at 7 and 30 days after treatment.
  The preoperative percussion values of the patient were marked on the visual analog scale by the patient. The intensity of the percussion was calculated by measuring the area in which the individual was marked between 0 (no pain) and 100 (severe pain). Patients recorded postoperative percussion levels on the VAS for pain from 0 (no pain) to 100 (worst pain) at 7 and 30 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Demet Altunbaş, DDS, PhD, Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas/Merkez, Turkey (Türkiye)

REFERENCES:
- [Derived] Ayhan M, Altunbas D. Efficacy of Potassium Titanyl Phosphate Laser and Sodium Hypochlorite on Postoperative Pain Intensity Following Pulpotomy in Teeth with Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial. Photobiomodul Photomed Laser Surg. 2023 May;41(5):225-233. doi: 10.1089/photob.2022.0152. Epub 2023 Apr 24. PMID 37092958